CLINICAL TRIAL: NCT01653327
Title: Analgesic Effects of Topical Ketamine Mouthwash in Patients Receiving Chemoradiation or Radiotherapy for Head and Neck Cancer
Brief Title: Analgesic Effects of Topical Ketamine Mouthwash in Patients Receiving Chemoradiation or Radiotherapy for Head & Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Thomas Davis, Staff Physician, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: D1022
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Results first posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Mucositis; Head and Neck Cancer
Keywords: mucositis; head and neck; cancer; radiation therapy; chemoradiation; oral; pain
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms; Neoplasms; Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Active Comparator): Twenty milligrams of ketamine will be dissolved in 4 mL of pharmaceutical cherry syrup and 1 ml of normal saline.
  Interventions: Drug: Ketamine
- Placebo (Placebo Comparator): The placebo will consist of 4 ml of cherry syrup and 1 ml of normal saline.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — Twenty milligrams of ketamine will be dissolved in 4 mL of pharmaceutical cherry syrup and 1 ml of normal saline.
  Arms: Ketamine
Drug: Placebo
  Arms: Placebo

SUMMARY:
* The primary objective is to determine the reduction in pain score by ketamine mouthwash compared to placebo in head and neck cancer patients with refractory mucositis.
* The secondary objectives are to describe the duration of analgesia and adverse effects associated with ketamine and placebo.

DETAILED DESCRIPTION:
We would like to determine the effectiveness of ketamine mouthwash in providing pain relief to subjects with head and neck cancer suffering from mucositis, a common adverse event of radiation therapy and chemoradiation therapy. Ketamine is a schedule III controlled substance that is generally used to provide anesthesia for short diagnostic and surgical procedures.

Ten subjects will be randomized to two treatment arms. Group A will receive ketamine on Monday, placebo on Wednesday, and ketamine on Friday. Group B will receive placebo on Monday, ketamine on Wednesday, and placebo on Friday. Each subject will swish the study drug or placebo for 2 minutes and spit it out. The use of non-maintenance mucositis medications such as DLM solution will not be allowed during the clinic visit. Subjects may resume non-maintenance mucositis medications at home.

Subjects will be asked to document adverse effects and pain scores at 30, 45, and 60 minutes after study medication. The Richmond Agitation and Sedation Scale (RASS) will be used to determine a subject's sedation level, if necessary. Treatment will last for up to 6 weeks unless an illness or an event occurs that prevents continuation, intolerance to the agent, adverse events, resolution of mucositis pain, or the decision to withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with head and neck tumors (any histology) receiving ongoing chemoradiation or radiation therapy
* Subjects with mucositis pain refractory to topical management, defined as any self-reported pain score of > 2 in the 24 hours prior to enrollment despite use of topical agents as prescribed
* Age ≥ 18 years
* Ability to understand and willingness to consent and to sign consent form

Exclusion Criteria:

* Active substance abuse at time of registration (alcohol, drugs, non-prescription use of controlled substances)
* Subjects with history of allergic reactions to ketamine
* Persistent oral bleeding: > 15 mL (estimated) per day
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-06; Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H David, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant recruitment occurred between 5/24/2010-8/3/2016.
Pre-assignment Details: Participants were randomized to receive ketamine (K) or placebo (P) in repeating sequences of KPK or PKP. Not all participants completed all sequences. A participant was considered complete if they received at least one dose of K or P and completed the pain assessment.
Groups:
- All Study Participants: Ketamine: Twenty milligrams of ketamine will be dissolved in 4 mL of pharmaceutical cherry syrup and 1 ml of normal saline.
  The placebo consisted of 4 ml of cherry syrup and 1 ml of normal saline.
Period: Overall Study
Arm/Group | All Study Participants
Started | 11
Completed (8 participants received both Ketamine and Placebo; 1 received Ketamine only; 2 received Placebo only) | 10
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort: All individuals participating in the trial.
Arm/Group | Cohort
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: Years] | 56.45 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Score
Description: The primary analysis is testing and estimating the effect of ketamine in comparison to placebo. Pain assessment will be analyzed using descriptive statistics. We will determine average pain scores. Pain will be measured using a 0-10 scale with 0 representing no pain; 1-3 representing mild pain; 4-6 representing moderate pain; and 7-10 representing severe pain. The effect of ketamine in comparison to placebo will be estimated with a mean and confidence interval. Proportional changes in pain scores (post-treatment pain score ÷ pre-treatment pain score) will be calculated and similarly analyzed. The proportion of subjects experiencing a reduction in pain scores of >33% will be calculated.
Time Frame: After 9-10 doses, expected average 1 month
Population: 1-4 pain measurements were obtained per participant. One assessment occurred per administered dose.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: Number of pain assessments
Groups:
- Placebo: The placebo consisted of 4 ml of cherry syrup and 1 ml of normal saline.
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 9 | 10
Number analyzed (Number of pain assessments) | 24 | 20
score on a scale | 1.167 (1.37) | 1.58 (1.31)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority; p = 0.3198, t-test, 2 sided

2. Secondary Outcome: Duration of Analgesic Effect
Description: The secondary analysis is testing and estimating the analgesic effect of ketamine in comparison to placebo. Pain assessment will be analyzed using descriptive statistics. We will also determine average duration of analgesia. The effect of ketamine in comparison to placebo will be estimated with a mean and confidence interval.
Time Frame: After 9-10 doses, expected average 1 month
Population: 1-4 measurements of analgesic effects were obtained per participant. One assessment occurred per administered dose.
Measure: Mean (Standard Deviation); unit: minutes
Units Other Than Participants: Total visits where duration was measured
Arm/Group | Ketamine | Placebo
Number analyzed (Participants) | 9 | 10
Number analyzed (Total visits where duration was measured) | 13 | 14
minutes | 39.231 (11.519) | 35.357 (9.499)
Statistical Analysis 1: Comparison: Ketamine vs Placebo; Test type: Superiority; p = 0.3522, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study, which is up to 6 weeks in total. For reporting purposes, if the adverse event occurred immediately after taking Ketamine or Placebo, the event is associated with that respective group.
Arm/Group | Ketamine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 3/9 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketamine (N=9) | Placebo (N=10)
Oral Pain; Grade 1 (General disorders) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes